CLINICAL TRIAL: NCT01257724
Title: Effects of an Evidence Service on Community-based AIDS Service Organizations' Use of Research Evidence: A Protocol for a Randomized Controlled Trial
Brief Title: Effects of an Evidence Service on Community-based AIDS Service Organizations' Use of Research Evidence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ontario HIV Treatment Network (Network)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Michael G. Wilson, Scientist, Health Policy & Knowledge Transfer and Exchange, Ontario HIV Treatment Network
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HHS/FHS REB 10-268
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Use of Research Evidence
Keywords: Knowledge translation; Community based organizations; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full-serve evidence service (Experimental): The full-serve evidence service consists of:
  1. an online searchable database of HIV-relevant systematic reviews;
  2. monthly email updates highlighting new reviews;
  3. access to user-friendly summaries produced by us or by others (when available);
  4. links to scientific abstracts;
  5. peer relevance assessments, which involves periodic requests to complete a brief assessment of how useful the information in the newly added review is with the average score posted once an assessment is completed;
  6. an interface for participants to leave comments in the records of systematic reviews in the database;
  7. links to full-text articles (when publicly available); and
  8. access to worksheets that help CBOs find and use research evidence
  Interventions: Other: SHARE (Synthesized HIV/AIDS Research Evidence)
- Self-serve evidence service (Active Comparator): Organizations allocated to the control group will only be provided website access to a listing of systematic reviews that are organized by year of publication with links to the record on PubMed (or another publicly available source when not available on PubMed) and access to worksheets that help community-based organizations find and use research evidence.
  Interventions: Other: SHARE (Synthesized HIV/AIDS Research Evidence)

INTERVENTIONS:
Other: SHARE (Synthesized HIV/AIDS Research Evidence) — SHARE (Synthesized HIV/AIDS Research Evidence) consists of several components:
  1. an online searchable database of HIV-relevant systematic reviews;
  2. monthly email updates highlighting new reviews;
  3. access to user-friendly summaries produced by us or by others (when available);
  4. links to scientific abstracts;
  5. peer relevance assessments, which involves periodic requests to complete a brief assessment of how useful the information in the newly added review is with the average score posted once an assessment is completed;
  6. an interface for participants to leave comments in the records of systematic reviews in the database;
  7. links to full-text articles (when publicly available); and
  8. access to worksheets that help CBOs find and use research evidence

SUMMARY:
The investigators have developed an online database called 'Synthesized HIV/AIDS Research Evidence' (SHARE), which is designed to support the use of research evidence by those working in the HIV/AIDS sector. This study will evaluate whether a "full-serve" version of SHARE increases the use of research evidence by community-based organizations as compared to a "self-serve" version. The "full-serve" version of SHARE consists of several components: 1) an online searchable database of synthesized research evidence relevant to HIV/AIDS , 2) periodic emailed updates, 3) access to user-friendly summaries and 4) peer-relevance assessments. The self-serve version consists only of a listing of relevant synthesized research evidence . The investigators will also interview participants in the study to obtain feedback about SHARE, how helpful it was in their work, why it was helpful (or not helpful), what aspects were most and least helpful and why, and recommendations for improving it.

DETAILED DESCRIPTION:
Background To support the use of research evidence by community-based organizations the investigators have developed 'Synthesized HIV/AIDS Research Evidence' (SHARE), which is an evidence service for those working in the HIV sector. SHARE consists of several components: 1) an online searchable database of HIV-relevant systematic reviews (retrievable based on a taxonomy of topics related to HIV/AIDS and open text search), 2) periodic email updates, 3) access to user-friendly summaries, and 4) peer relevance assessments. The objective is to evaluate whether this "full serve" evidence service increases the use of research evidence by community-based organizations as compared to a "self-serve" evidence service.

Methods/design The investigators will conduct a two-arm randomized controlled trial (RCT), along with a follow-up qualitative process study to explore the findings in greater depth. All community-based organizations affiliated with Canadian AIDS Society (n=120) will be invited to participate and will be randomized to receive either the "full-serve" version of SHARE or the "self-serve" version (a listing of relevant systematic reviews with links to records on PubMed and worksheets that help community-based organizations find and use research evidence) using a simple randomized design. All management and staff from each organization will be provided access to the version of SHARE that their organization is allocated to. The trial duration will be 10 months (two-month baseline period, six-month intervention period, and two month cross-over period), the primary outcome measure will be the mean number of logins/month/organization (averaged across the number of users from each organization) between baseline and the end of the intervention period and the secondary outcome will be intention to use research evidence as measured by a survey administered to one key decision-maker from each organization. For the qualitative study, one key organizational decision-maker from 15 organizations in each trial arm (n=30) will be purposively sampled. One-on-one semi-structured interviews will be conducted by telephone on their views about and their experiences with the evidence service they received, how helpful it was in their work, why it was helpful (or not helpful), what aspects were most and least helpful and why, and recommendations for next steps.

ELIGIBILITY:
Inclusion Criteria:

* We will include all community-based organizations affiliated with the Canadian AIDS Society and from relevant provincial HIV/AIDS networks in Canada.

Exclusion Criteria:

* We will exclude organizations that do not have at least one key decision-maker who is comfortable participating and corresponding in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
number of logins/month/organization | 6 months
  The investigators will track utilization of the evidence service at the organizational level by calculating the mean number of logins/month/organization (the total organizational logins/month will be averaged across the number of users from each organization).

SECONDARY OUTCOMES:
Intention to use research evidence | Baseline and follow-up (after delivery of 6-month intervnetion)
  The investigators will use the theory of planned behaviour to measure participants' intention to use research. Using a manual designed to construct measures based on the theory, colleagues have developed and sought preliminary feedback on a data-collection instrument by first assessing face validity through interviews with key informants and then pilot testing it with 28 policymakers and researchers who completed it after participating in a knowledge translation intervention. In addition, colleagues found the data-collection instrument to have moderate test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Wilson, PhD, Principal Investigator — McMaster University; Ontario HIV Treatment Network; John N Lavis, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Ontario HIV Treatment Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wilson MG, Lavis JN, Grimshaw JM, Haynes RB, Bekele T, Rourke SB. Effects of an evidence service on community-based AIDS service organizations' use of research evidence: a protocol for a randomized controlled trial. Implement Sci. 2011 May 27;6:52. doi: 10.1186/1748-5908-6-52. PMID 21619622